CLINICAL TRIAL: NCT05737251
Title: Positive Emotions Training (PoET) as an Online Intervention to Improve Mental Health: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Lara Niemann, Master of Science (M.Sc.) in Clinical Psychology, Ruhr University of Bochum
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PoET101
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Positive Emotions; Mental Health
Keywords: positive emotions; online intervention; positive psychology
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PoET Group (Experimental): Participants received two sessions of PoET and filled out the questionnaires.
  Interventions: Behavioral: PoET
- Control Group (No Intervention): Participants only filled out the questionnaires.

INTERVENTIONS:
Behavioral: PoET — PoET consists of two online-sessions, each 3.5 hours within groups of 30 people. The following lessons regarding positive psychology constructs were conducted (including short information on each construct and specific exercises): happiness, hope, humour, optimism, gratitude, self-efficacy, flow, meaningfulness, forgiveness, spirituality and resilience.
  Arms: PoET Group

SUMMARY:
Positive psychology interventions are known to have an impact on mental health as well as on a number of beneficial characteristics like optimism, gratitude and self-efficacy. The new developed Positive Emotions Training (PoET) is one of the first holistic training programs covering eleven positive psychology constructs. The goal of this study was to test PoET's feasibility in the general population and to assess possible effects on positive and negative mental health factors. Additionally, possible effects on optimism, gratitude, happiness, resilience, and self-efficacy were examined.

Hypotheses:

1. It was hypothesized that participants receiving PoET would show a significant increase in positive mental health factors one month after the second training day.
2. It was expected to find a significant decrease in depression, anxiety, and stress symptoms one month after the second training day.
3. It was hypothesized that participants in a control group would not show any significant changes in this regard.

Methods:

The sample (n = 101) was allocated to PoET (n = 55) or control (n = 46) which did not receive any treatment. The allocation was neither randomized nor matched. Participants in the PoET group completed a whole of two training sessions (3.5 hours each) that were conducted in an online format (via Zoom) with groups of about 30 people. These sessions included the following positive psychology constructs: happiness, hope, humour, optimism, gratitude, self-efficacy, flow, meaningfulness, forgiveness, spirituality, resilience.

All participants completed positive and negative mental health measures at the beginning of the first training session and at the beginning of the second one as well as 30 days after the second session. Additionally, they had to complete two short items regarding stress and mood after each training session. They were given an exercise booklet with descriptions and explanations for all exercises during the training and at home. The week between the two sessions was called "7-day-challenge" to motivate the participants to try out several exercises at home.

Data was collected pseudonymised via Socisurvey. Data analysis was conducted with RStudio. Two-factorial repeated measures ANOVAs were conducted to test for possible effects of PoET on mental health.

ELIGIBILITY:
Inclusion Criteria:

* legal age (18)
* ability to use Zoom and all associated technology

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in Positive Mental Health Scale (3 assessment points) | before 1st and 2nd training session, 30 days after 2nd training session
  9 items, 4-point-scale from 0 ("I do not agree ") to 3 ("I agree"), assessing emotional and psychological aspects of wellbeing, higher scores reflect better positive mental health
Changes in Depression Anxiety Stress Scale 21 (3 assessment points) | before 1st and 2nd training session, 30 days after 2nd training session
  21 items, 4-point-scale from 0 ("did not apply to me at all") to 3 ("applied to me very much or most of the time"), assessing negative emotional states, higher scores reflect more symptoms of depression, anxiety and stress

SECONDARY OUTCOMES:
Changes in Life Orientation Test-revised (3 assessment points) | before 1st and 2nd training session, 30 days after 2nd training session
  10 items, 5-point-scale from 0 ("strongly disagree") to 4 ("strongly agree"), assessing dispositional optimism, higher scores reflect higher dispositional optimism
Changes in Gratitude Questionnaire (3 assessment points) | before 1st and 2nd training session, 30 days after 2nd training session
  5 items, 7-point-scale from 1 ("strongly disagree") to 7 ("strongly agree"), assessing gratitude, higher scores reflect a more pronounced sense of gratitude
Changes in Satisfaction With Life Scale (3 assessment points) | before 1st and 2nd training session, 30 days after 2nd training session
  5 items, 7-point-scale from 1 ("strongly disagree") to 7 ("strongly agree"), assessing global subjective happiness, higher scores indicate a happier person
Changes in New General Self-Efficacy Scale (3 assessment points) | before 1st and 2nd training session, 30 days after 2nd training session
  8 items, 5-point-scale from 1 ("strongly disagree") to 5 ("strongly agree"), assessing how much participants believe in their own abilities, higher scores represent higher self-efficacy
Changes in Brief Resilience Scale (3 assessment points) | before 1st and 2nd training session, 30 days after 2nd training session
  6 items, 5-point-scale from 1 ("strongly disagree") to 5 ("strongly agree"), assessing participants' ability to recover from stress despite significant adversity, higher scores reflect higher resilience

CONTACTS AND LOCATIONS:
Overall Officials: Christina Totzeck, Dr., Study Director — Ruhr-University Bochum
Locations (1):
- Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niemann L, von Gruner C, Zhang XC, Margraf J, Totzeck C. Positive Emotions Training (PoET) as an online intervention to improve mental health: a feasibility study. BMC Public Health. 2023 Aug 14;23(1):1543. doi: 10.1186/s12889-023-16424-x. PMID 37580658